CLINICAL TRIAL: NCT06247943
Title: Lung Protective Ventilation Strategies to Improve Oxygenation Function and Respiratory Mechanics in Patients Undergoing Robotic Bariatric Surgery
Brief Title: Lung Protective Ventilation Strategies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin Medical University General Hospital (Other)
Responsible Party: Principal Investigator, Guolin Wang, professor, Tianjin Medical University General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: GWang026
Record Dates: First submitted 2023-12-25; First posted 2024-02-08 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Respiration
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lung Protective Ventilation Strategy Group (Experimental): Use of lung-protective ventilation strategies
  Interventions: Procedure: Lung Protective Ventilation Strategy
- Control Group (Other): Use of general ventilation strategies
  Interventions: Procedure: regular ventilation

INTERVENTIONS:
Procedure: Lung Protective Ventilation Strategy — After 10 minutes of pneumoperitoneum, VT 7 ml/kg was used, PEEP 6 cmH2O, FiO2 was 40%, and plateau pressure <30 cmH2O was maintained throughout.
  Arms: Lung Protective Ventilation Strategy Group
Procedure: regular ventilation — VT 9ml /kg without PEEP, FiO2 of 60%
  Arms: Control Group

SUMMARY:
Obesity is becoming a common condition and bariatric metabolic surgery is one of the main options for treating morbid obesity. However, since most patients undergoing robotic bariatric surgery are class III obese, it brings new challenges to perioperative anesthesia management. Here, we explored the effects of lung-protective ventilation strategies on pulmonary oxygenation function and respiratory mechanics in patients undergoing robotic bariatric surgery.

DETAILED DESCRIPTION:
Forty obese patients who underwent robotic bariatric surgery in our hospital were selected and randomly divided into a lung-protective ventilation strategy group (Group P) and a control group (Group C). The volume-controlled mode was used to assist ventilation, and the inspiratory/expiratory ratio (I: E) was 1:2. Tidal volume (VT) was set according to the Predicted body weight (PBW) throughout the whole procedure, and in group C, VT was 9 ml /kg without Positive end-expiratory pressure (PEEP), and the inhaled oxygen concentration (Fraction of oxygen) was 0.5 ml /kg, while the inspiratory oxygen concentration (Fraction of oxygen) was 0.5 ml /kg. Group C: VT 9ml /kg, no Positive end-expiratory pressure (PEEP), Fraction of inspiration O2 (FiO2) of 60%; Group P: the ventilation mode was the same as that of Group C from tracheal intubation to the beginning of pneumoperitoneum for 10 minutes, and after 10 minutes of pneumoperitoneum, the ventilation mode was the same as that of Group C. After the pneumoperitoneum for 10 minutes, the ventilation mode was VT 7ml/kg, PEEP 6cmH2O, FiO2 of 40%, and the plateau pressure was maintained at <30cmH2O. In both groups, the intraoperative gas flow was 2L/min, and SpO2 was maintained at ≥95%; if it could not be maintained, the oxygenation function of the patients could be improved by adjusting the ventilation parameters and strategies; meanwhile, the respiratory rate (RR) was adjusted to maintain the End-tidal carbon dioxide partial pressure (PETCO2) at ≥30%, and the end-tidal carbon dioxide partial pressure (PETCO2) was maintained at ≥30%, and the end-tidal carbon dioxide partial pressure (PETCO2) was maintained at ≥30%. The respiratory mechanical parameters: tidal volume, RR, airway peak pressure (PPeak), plateau pressure (PPeak), and plateau pressure (PPeak) were recorded at 5 minutes after tracheal intubation (T0), 10 minutes after the start of the pneumoperitoneum (T1), 60 minutes (T2), 120 minutes (T3), and 10 minutes after the pneumoperitoneum was closed (T4). pressure (PPeak), and plateau pressure (PPlate), and calculate the dynamic lung compliance; arterial blood was drawn at T0, T1, T2, T3, and T4, respectively, and the arterial partial pressure of oxygen (PaO2) and the arterial partial pressure of carbon dioxide (Arterial CO2) were measured. The arterial partial pressure of oxygen (PaO2) and arterial carbon dioxide pressure (PaCO2) were measured, and the oxygenation index (OI) was calculated.

ELIGIBILITY:
Inclusion Criteria:

Obese patients with ASA grade Ⅰ ~ Ⅲ No obvious abnormality in preoperative lung function and blood gas analysis results Undergoing robotic bariatric surgery

Exclusion Criteria:

Had been mechanically ventilated 2 weeks before surgery Thoracic deformity Neuromuscular disease Significant abnormalities in vital organ function Combined pneumothorax or pulmonary herniation Participating in other clinical intervention trials or refusing general anesthesia with tracheal intubation Emergency surgery

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-03-16 (Actual); Study Completion 2024-03-17 (Actual)

PRIMARY OUTCOMES:
Respiratory mechanics | 5 minutes after tracheal intubation (T0), 10 minutes after the start of pneumoperitoneum (T1), 60 minutes (T2), 120 minutes (T3), and 10 minutes after the closure of the pneumoperitoneum (T4)
  plateau airway pressure
oxygenation | 5 minutes after tracheal intubation (T0), 10 minutes after the start of pneumoperitoneum (T1), 60 minutes (T2), 120 minutes (T3), and 10 minutes after the closure of the pneumoperitoneum (T4)
  Oxygenation index
oxygenation | 5 minutes after tracheal intubation (T0), 10 minutes after the start of pneumoperitoneum (T1), 60 minutes (T2), 120 minutes (T3), and 10 minutes after the closure of the pneumoperitoneum (T4)
  arterial oxygen partial pressure
Respiratory mechanics | 5 minutes after tracheal intubation (T0), 10 minutes after the start of pneumoperitoneum (T1), 60 minutes (T2), 120 minutes (T3), and 10 minutes after the closure of the pneumoperitoneum (T4)
  peak airway pressure
Respiratory mechanics | 5 minutes after tracheal intubation (T0), 10 minutes after the start of pneumoperitoneum (T1), 60 minutes (T2), 120 minutes (T3), and 10 minutes after the closure of the pneumoperitoneum (T4)
  end-tidal carbon dioxide partial pressure

SECONDARY OUTCOMES:
Hemodynamics | 5 minutes after tracheal intubation (T0), 10 minutes after the start of pneumoperitoneum (T1), 60 minutes (T2), 120 minutes (T3), and 10 minutes after the closure of the pneumoperitoneum (T4)
  mean arterial pressure
complications | postoperative days 1, 3, and 5
  postoperative pulmonary complications

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University General Hospital, Tianjin, China